CLINICAL TRIAL: NCT03070769
Title: Evaluation of Inflammatory Markers in a Large Sample of Obstructive Sleep Apnea Patients
Brief Title: Inflammatory Markers in Obstructive Sleep Apnea (OSA) Patients.
Status: Completed | Type: Observational
Sponsor: University of Crete (Other)
Responsible Party: Principal Investigator, Izolde Bouloukaki, Principal Investigator, University of Crete
Other Study IDs: OSAINFL1
Record Dates: First submitted 2017-02-24; First posted 2017-03-06 (Actual); Last update posted 2017-03-06 (Actual); Status verified 2017-03

CONDITIONS: Obstructive Sleep Apnea of Adult

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Subjects without Obstructive sleep apnea (Apnea-hypopnea index-AHI<5). Venous blood collection for biomarkers measurements.
  Interventions: Procedure: Venous blood collection for biomarkers measurements
- Obstructive sleep apnea (OSA) patients: Patients with Obstructive sleep apnea (AHI> or =5). Venous blood collection for biomarkers measurements.
  Interventions: Procedure: Venous blood collection for biomarkers measurements

INTERVENTIONS:
Procedure: Venous blood collection for biomarkers measurements — Venous blood was collected in all subjects for measurements of hs-C-reactive protein (hs-CRP), fibrinogen, erythrocyte sedimentation rate (ESR) and Uric Acid (UA) between 8:00 and 9:00 AM, following an overnight fast, shortly after the conclusion of the overnight polysomnography (PSG).

SUMMARY:
The aim of our study was to assess the levels of inflammatory biomarkers in a large sample of OSA patients and to investigate any correlation between these markers with clinical and polysomnographic (PSG) parameters.

Subjects undergone a PSG for OSA diagnosis were recruited. Patients with known comorbidities were excluded from the study. Included patients were grouped according to apnea-hypopnea index (AHI) as mild, moderate and severe. Patients with AHI < 5 served as control group. Demographic, PSG data, serum levels of hs-C-reactive protein (hs-CRP), fibrinogen, erythrocyte sedimentation rate (ESR) and Uric Acid (UA) were measured and compared between groups.

DETAILED DESCRIPTION:
Systemic inflammation is important in obstructive sleep apnea (OSA) pathophysiology and its comorbidity. The objective of this study was to investigate how early biomarkers of inflammation may be altered in OSA patients. To complete this goal the investigators assessed the circulating levels of four inflammatory markers, hs-C-reactive protein (hs-CRP), Fibrinogen, erythrocyte sedimentation rate (ESR) and Uric Acid (UA) in a representative population of consecutively enrolled, untreated and otherwise healthy subjects with a clinical suspicion of obstructive sleep apnea. A secondary objective was to investigate any correlation between these markers with clinical and polysomnographic (PSG) parameters of these subjects.Subjects who had undergone a PSG for OSA diagnosis were recruited. Patients with known comorbidities were excluded from the study. Included patients were grouped according to apnea-hypopnea index (AHI) as mild, moderate and severe. Patients with AHI < 5 served as control group. Demographic, PSG data, serum levels of hs-CRP, fibrinogen, ESR and UA were measured and compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed, untreated, and otherwise healthy obstructive sleep apnea (OSA) patients
* healthy subjects (without OSA)

Exclusion Criteria:

* refusal to participate,
* previous OSA diagnosis and treatment
* known comorbidities,
* pregnancy,
* history of narcolepsy or restless leg syndrome.
* Subjects younger than 18 years,
* Central sleep apnea syndrome (CSAS) diagnosed with PSG,

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consecutive patients, who were admitted to the Sleep Disorders Center, Department of Thoracic Medicine, University of Crete Medical School, for evaluation of suspected sleep-disordered breathing, were considered as potential recruits for this study.
Sampling Method: Probability Sample
Enrollment: 1053 (Actual)
Dates: Start 2012-06-01 (Actual); Primary Completion 2016-06-01 (Actual); Study Completion 2016-12-12 (Actual)

PRIMARY OUTCOMES:
Inflammatory biomarkers levels in OSA patients without comorbidities compared to controls. | 4 years
  Inflammatory biomarkers levels in OSA patients without comorbidities compared to controls,as assessed by high sensitive -C-reactive protein (hs-CRP), Fibrinogen, Erythrocyte sedimentation rate (ESR) and uric acid (UA).

CONTACTS AND LOCATIONS:
Overall Officials: Sophia Schiza, MD, PhD, Study Chair — University of Crete
Locations (1):
- Sleep Disorders Center, Department of Thoracic Medicine, University of Crete,, Heraklion, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bouloukaki I, Mermigkis C, Tzanakis N, Kallergis E, Moniaki V, Mauroudi E, Schiza SE. Evaluation of Inflammatory Markers in a Large Sample of Obstructive Sleep Apnea Patients without Comorbidities. Mediators Inflamm. 2017;2017:4573756. doi: 10.1155/2017/4573756. Epub 2017 Jul 31. PMID 28831208